CLINICAL TRIAL: NCT02582801
Title: 18F-Alfatide Ⅱ PET/CT in the Diagnosis and Treatment Response Evaluation of Breast Cancer Patients
Brief Title: Clinical Research of 18F-Alfatide Ⅱ PET/CT in Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The cyclotron in our hospital has a serious malfunction and can not be repaired. It will take a long time to purchase and install the new cyclotron.
Sponsor: Jiang Wu (Other)
Responsible Party: Sponsor-Investigator, Jiang Wu, Medical doctor, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Molecular Imaging
Record Dates: First submitted 2015-10-20; First posted 2015-10-21 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer
Keywords: PET/CT; Alfatide Ⅱ; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — alfatide II

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- breast cancer (Experimental): Perform 18F-Alfatide Ⅱ PET/CT in breast cancer patients
  Interventions: Drug: 18F-Alfatide Ⅱ PET/CT
- benign breast lesions (Active Comparator): Perform 18F-Alfatide Ⅱ PET/CT in patients with benign breast lesions
  Interventions: Drug: 18F-Alfatide Ⅱ PET/CT

INTERVENTIONS:
Drug: 18F-Alfatide Ⅱ PET/CT — Inject 18F-Alfatide Ⅱ by vein and then perform PET/CT scan after 60 min
  Other Names: 18F-AlF-NOTA-E[PEG4-c(RGDfk)]2

SUMMARY:
18F-Alfatide Ⅱ PET/CT in breast cancer patients

DETAILED DESCRIPTION:
The investigators aim to assess the clinical application of 18F-Alfatide Ⅱ PET/CT in the diagnosis and treatment response monitoring of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patients have been suspected or diagnosed with breast cancer and they have not received any treatment; It must fulfill the ethical requirements and subjects have signed an informed consent.

Exclusion Criteria:

* Pregnancy or nursing mothers; Those patients accompanied by other serious diseases such as cardiac functional insufficiency, hepatic and renal function insufficiency.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Maximum standardized uptake value (SUVmax) | 1 day
  the uptake intensity of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Guangming Lu, Professor, Study Chair — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yu C, Pan D, Mi B, Xu Y, Lang L, Niu G, Yang M, Wan W, Chen X. (18)F-Alfatide II PET/CT in healthy human volunteers and patients with brain metastases. Eur J Nucl Med Mol Imaging. 2015 Dec;42(13):2021-8. doi: 10.1007/s00259-015-3118-2. Epub 2015 Jul 1. PMID 26121930
- [Background] Wang SY, Bao X, Wang MW, Zhang YP, Zhang YJ, Zhang JP. Radiation dosimetry estimates of (18)F-alfatide II based on whole-body PET imaging of mice. Appl Radiat Isot. 2015 Nov;105:1-5. doi: 10.1016/j.apradiso.2015.07.013. Epub 2015 Jul 13. PMID 26218449
- [Background] Mi B, Yu C, Pan D, Yang M, Wan W, Niu G, Chen X. Pilot Prospective Evaluation of (18)F-Alfatide II for Detection of Skeletal Metastases. Theranostics. 2015 Jul 12;5(10):1115-21. doi: 10.7150/thno.12938. eCollection 2015. PMID 26199649
- [Background] Wu C, Yue X, Lang L, Kiesewetter DO, Li F, Zhu Z, Niu G, Chen X. Longitudinal PET imaging of muscular inflammation using 18F-DPA-714 and 18F-Alfatide II and differentiation with tumors. Theranostics. 2014 Feb 26;4(5):546-55. doi: 10.7150/thno.8159. eCollection 2014. PMID 24672585
- [Background] Guo J, Guo N, Lang L, Kiesewetter DO, Xie Q, Li Q, Eden HS, Niu G, Chen X. (18)F-alfatide II and (18)F-FDG dual-tracer dynamic PET for parametric, early prediction of tumor response to therapy. J Nucl Med. 2014 Jan;55(1):154-60. doi: 10.2967/jnumed.113.122069. Epub 2013 Nov 14. PMID 24232871